CLINICAL TRIAL: NCT04388215
Title: A Randomized, Double-blind, Multi-center, Therapeutic Confirmatory, Phase 3 Trial to Evaluate the Efficacy and Safety of CKD-828, D326, and D337 Combination Therapy in Hypertensive Patients With Dyslipidemia
Brief Title: Clinical Study to Evaluate the Efficacy and Safety of CKD-348(CKD-828, D326, D337) Tablet
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A86_03HT/DL1905
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Hypertension; Dyslipidemias
MeSH Terms: conditions — Hypertension; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group (Experimental): Drug: CKD-828 80/5mg, D326 20mg, D337 10mg, D013(placebo) 80mg
  - CKD-828 80/5mg, D326 20mg, D337 10mg, D013(placebo) 80mg, orally, 1 tablet once a day for 8 weeks
  Interventions: Drug: CKD-828; Drug: D326; Drug: D337; Drug: D013(placebo)
- Comparator group 1 (Active Comparator): Drug: CKD-828 80/5mg, D326(placebo) 20mg, D337(placebo) 10mg, D013(placebo) 80mg
  - CKD-828 80/5mg, D326(placebo) 20mg, D337(placebo) 10mg, D337(placebo) 10mg, D013(placebo) 80mg, orally, 1 tablet once a day for 8 weeks
  Interventions: Drug: CKD-828; Drug: D326(placebo); Drug: D337(placebo); Drug: D013(placebo)
- Comparator group 2 (Active Comparator): Drug: CKD-828(placebo) 80/5mg, D326 20mg, D337 10mg, D013 80mg
  - CKD-828(placebo) 80/5mg, D326 20mg, D337 10mg, D013 80mg, orally, 1 tablet once a day for 8 weeks
  Interventions: Drug: CKD-828(placebo); Drug: D326; Drug: D337; Drug: D013

INTERVENTIONS:
Drug: CKD-828 — orally, 1 tablet once a day for 8 weeks
  Arms: Comparator group 1; Treatment group
Drug: CKD-828(placebo) — orally, 1 tablet once a day for 8 weeks
  Arms: Comparator group 2
Drug: D326 — orally, 1 tablet once a day for 8 weeks
  Arms: Comparator group 2; Treatment group
Drug: D326(placebo) — orally, 1 tablet once a day for 8 weeks
  Arms: Comparator group 1
Drug: D337 — orally, 1 tablet once a day for 8 weeks
  Arms: Comparator group 2; Treatment group
Drug: D337(placebo) — orally, 1 tablet once a day for 8 weeks
  Arms: Comparator group 1
Drug: D013 — orally, 1 tablet once a day for 8 weeks
  Arms: Comparator group 2
Drug: D013(placebo) — orally, 1 tablet once a day for 8 weeks
  Arms: Comparator group 1; Treatment group

SUMMARY:
to evaluate the efficacy and safety of CKD-828, D326, and D337 combination therapy in Hypertensive patients with Dyslipidemia

DETAILED DESCRIPTION:
The purpose of this phase III study was to evaluate the efficacy and safety of CKD-348(CKD-828, D326, D337) tablet administration for treatment period(8 weeks) in essential hypertesive patients with Dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

1. Between 19 years and 75 years old(male or female)
2. Diagnosed essential hypertensive patients with dyslipidemia or the patients who has been taking antihypertensive and antidyslipidemic drugs
3. The patients who can stop taking antihypertensive and antidyslipidemic drugs accroding to Principle Investigator's opinion
4. Agreement with written informed consent

Exclusion Criteria:

1. Patients whose blood pressure measured at screening is one of the following:

   * Mean Sitting Systolic Blood Pressure ≥ 200 mmHg or Mean Sitting Diastolic Blood Pressure ≥ 120 mmHg
   * Difference in Mean Sitting Systolic Blood Pressure between patient's both arms ≥ 20 mmHg and Mean Sitting Diastolic Blood Pressure ≥ 10 mmHg
2. Patients whose lipid level measured at screening is one of the following:

   * Low Density Lipoprotein-C > 250 mg/dL or Triglyceride ≥ 500 mg/dL
3. Patients diagnosed with secondary hypertension or suspected of secondary hypertension(coarctation of aorta, primary aldosteronism, etc).

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-10-23 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Change rate from baseline in Low Density Lipoprotein-C | Baseline, 8 weeks
  (compare treatment group with comparator group 1)
Change from baseline in Mean Sitting Systolic Blood Pressure | Baseline, 8 weeks
  (compare treatment group with comparator group 2)

SECONDARY OUTCOMES:
Change rate from baseline in Low Density Lipoprotein-C | Baseline, 4 weeks
Change from baseline in Low Density Lipoprotein-C | Baseline, 4 weeks, 8 weeks
Change and change rate from baseline in Total Cholesterol, Triglyceride, High Density Lipoprotein-C | Baseline, 4 weeks, 8 weeks
Low Density Lipoprotein-C target achievement rate accroding to National Cholesterol Education Program(NCEP) Third Adult Treatment Panel(ATP III) guideline at 4 weeks and 8 weeks | Baseline, 4 weeks, 8 weeks
Change from baseline in Mean Sitting Systolic Blood Pressure | Baseline, 4 weeks
Change from baseline in Mean Sitting Diastolic Blood Pressure | Baseline, 4 weeks, 8 weeks
Normalization rate of blood pressure after 4 weeks and 8 weeks | Baseline, 4 weeks, 8 weeks
  Blood Pressure < 140/90 mmHg

OTHER OUTCOMES:
Change and change rate from baseline in Low Density Lipoprotein-C, Total Cholesterol, Triglyceride, High Density Lipoprotein-C | Baseline, 4 weeks, 8 weeks
Low Density Lipoprotein-C target achievement rate accroding to National Cholesterol Education Program(NCEP) Third Adult Treatment Panel(ATP III) guideline at 4 weeks and 8 weeks | Baseline, 4 weeks, 8 weeks
Change from baseline in Mean Sitting Systolic Blood Pressure and Mean Mean Sitting Diastolic Blood Pressure | Baseline, 4 weeks, 8 weeks
Normalization rate of blood pressure after 4 weeks and 8 weeks | Baseline, 4 weeks, 8 weeks
  Blood Pressure < 140/90 mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No